CLINICAL TRIAL: NCT06160622
Title: A Phase I Single Dose, Non-Randomised, Open-Label, Parallel Group Study to Investigate the Effect of Severe Kidney Impairment on the Pharmacokinetics, Safety and Tolerability of Leritrelvir(RAY1216)
Brief Title: Pharmacokinetics of Leritrelvir(RAY1216) in Participants With Severe Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RAY1216-23-07
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Kidney Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental 1: participants with severe renal impairment (Experimental): 8 participants with severe renal impairment will be given 400mg of Leritrelvir
  Interventions: Drug: Leritrelvir
- Experimental 2: healthy participants (Experimental): 8 participants with normal renal function will be given 400mg of Leritrelvir
  Interventions: Drug: Leritrelvir

INTERVENTIONS:
Drug: Leritrelvir — Oral

SUMMARY:
This study will assess the effect of severe kidney impairment on the pharmacokinetics (PK), safety and tolerability of Leritrelvir.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥19 to ≤28kg/m2 and total body weight >50 kg(male) or >40kg(female) at Screening (calculated as a function of measured height and weight according to the formula, BMI = kg / m2 where m2 is height in meters squared);
2. Ability to understand and willingness to sign a written informed consent form;

   Participants with normal renal function only:
3. Normal physical examination, vital signs, 12-lead ECG, Chest X-ray images (anteroposterior) and clinical laboratory values, or any abnormality that is non-clinically significant.
4. Glomerular filtration rate (GFR)≥ 90 mL/min
5. Age, BMI, and sex comparable to those of subjects of severe renal impairment

   Participants with severe renal impairment only:
6. Diagnosis of CKD at least 3 months
7. glomerular filtration rate (GFR)< 60 mL/min/1.73 m2

Exclusion Criteria:

1. Participants with an allergic disposition (multiple drug and food allergies) or who, as determined by the investigator, are likely to be allergic to the investigational drug product or any component of the investigational drug product.
2. Participants who donated blood or bleeding profusely (> 400 mL) in the 3 months.
3. Pregnant or lactating women, or women of childbearing age with a positive pregnancy test
4. Participants with serious infections, trauma, gastrointestinal surgery or other major surgical procedures within 4 weeks

   Participants with severe renal impairment only:
5. Participants with acute renal failure, or a kidney transplant history; Or requiring renal dialysis during the study period;
6. Hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥ 160mm Hg or diastolic blood pressure ≥ 100mm)
7. New York heart association (NYHA) class III or IV congestive heart failure
8. Alanine aminotransferase (ALT) ≥ 2×ULN, aspartate aminotransferase(AST) ≥ 2×ULN; Serum total bilirubin > 1.5×ULN;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 0~96 hours
  The Cmax of a single dose of Leritrelvir in participants with severe impaired renal function and controls with normal renal function will be evaluated and compared.
Area under the concentration-time curve from time zero to last time of quantifiable concentration (AUClast) | 0~96 hours
  The AUClast of a single dose of Leritrelvir in participants with severe impaired renal function and controls with normal renal function will be evaluated and compared.

SECONDARY OUTCOMES:
Number of participants with drug-related adverse events as assessed by CTCAE v5.0 | Day 1 to Day12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China